CLINICAL TRIAL: NCT04799249
Title: A Phase 3, Randomized, Double-Blind Study of Trilaciclib or Placebo in Patients Receiving First- or Second-Line Gemcitabine and Carboplatin Chemotherapy for Locally Advanced Unresectable or Metastatic Triple-Negative Breast Cancer (PRESERVE 2)
Brief Title: Trilaciclib, a CDK 4/6 Inhibitor, in Patients Receiving Gemcitabine and Carboplatin for Metastatic Triple-Negative Breast Cancer (TNBC)
Acronym: PRESERVE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G1T28-208; 2020-004930-39 (EudraCT Number)
Record Dates: First submitted 2021-02-18; First posted 2021-03-16 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: TNBC - Triple-Negative Breast Cancer; Breast Cancer
Keywords: breast cancer; gemcitabine; carboplatin; solid tumors; breast; chemotherapy; TNBC; trilaciclib; cyclin-dependent kinase 4/6 inhibitor; CDK 4/6 Inhibitor; triple-negative breast cancer; metastatic; chemotherapy-induced fatigue; HER2-negative; immunotherapy; immune checkpoint inhibitor therapy; chemotherapy-induced myelosuppression; myeloprotection; myeloprotective; PD-1/PD-L1 inhibitor therapy; advanced; stage 4; preserve; PRESERVE 2
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms; Neoplasm Metastasis | interventions — trilaciclib; Saline Solution; Glucose; Water; Gemcitabine; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trilaciclib + gemcitabine + carboplatin (Experimental): Trilaciclib (240mg/m2) + gemcitabine (1000 mg/m2) and carboplatin (AUC 2)
  Interventions: Drug: Trilaciclib; Drug: Gemcitabine; Drug: Carboplatin
- Placebo + gemcitabine + carboplatin (Placebo Comparator): The subjects in the placebo arm will follow the same schedule as the trilaciclib arm, but will receive placebo instead of trilaciclib.
  Interventions: Drug: Placebo; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Trilaciclib — Trilaciclib administered IV over 30mins prior to chemotherapy on Day 1 and Day 8 of each 21-day cycle.
  Other Names: G1T28; COSELA
  Arms: Trilaciclib + gemcitabine + carboplatin
Drug: Placebo — Placebo administered IV over 30mins prior to chemotherapy on Day 1 and Day 8 of each 21-day cycle.
  Other Names: 0.9% normal saline; 5 % Dextrose in water (D5W)
  Arms: Placebo + gemcitabine + carboplatin
Drug: Gemcitabine — Gemcitabine administered IV on Day 1 and Day 8 of each 21-day cycle.
Drug: Carboplatin — Carboplatin administered IV on Day 1 and Day 8 of each 21-day cycle.

SUMMARY:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled study evaluating the safety and efficacy of trilaciclib versus placebo administered prior to gemcitabine and carboplatin in patients receiving first- or second-line treatment for locally advanced unresectable/metastatic TNBC.

DETAILED DESCRIPTION:
This study will have two separate cohorts (Cohort 1 and Cohort 2). Both cohorts will follow the same general study conduct/design with similar primary and key secondary endpoints and identical treatment arms.

* Cohort 1 will evaluate patients receiving first-line therapy, regardless of programmed death-ligand 1 (PD-L1) status, who are programmed cell death protein 1 (PD-1)/PD-L1 inhibitor therapy naïve.
* Cohort 2 will evaluate PD-L1 positive patients receiving second-line therapy following prior PD-1/PD-L1 inhibitor therapy in the locally advanced unresectable/metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Age >/= 18 years of age with evaluable locally advanced unresectable or metastatic TNBC.
2. Documentation of triple negative breast cancer (estrogen and progesterone receptor <1% and HER2-negative)
3. Prior systemic therapies (Cohort 1 only):

   1. No prior systemic therapy in the locally advanced unresectable/metastatic setting including chemotherapy, targeted therapy, immunotherapy, or investigational agents.
   2. Prior PD-1/PD-L1 inhibitor treatment is not permitted in any setting, including in the neoadjuvant setting.
   3. Time between completion of last treatment with curative intent and first metastatic recurrence must be ≥ 6 months.
4. Prior systemic therapies (Cohort 2 only):

   1. Documentation of PD-L1 positive status
   2. Treated with a PD-1/PD-L1 inhibitor for a minimum duration of 4 months in the locally advanced unresectable/metastatic setting and as the most recent therapy.
5. Radiation therapy for metastatic disease is permitted. There is no required minimum washout period for radiation therapy. Patients should be recovered from the effects of radiation.
6. Archival tumor tissue must be available or a fresh biopsy must be obtained, unless approved by the Medical Monitor.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
8. Adequate organ function as demonstrated by normal laboratory values

Exclusion Criteria:

1. Prior treatment with gemcitabine in any setting.
2. Prior treatment with carboplatin in the locally advanced unresectable/metastatic setting.

   Prior carboplatin in the (neo)adjuvant/curative setting is permitted as long as it was completed ≥ 6 months prior to the first metastatic recurrence.
3. Presence of central nervous system (CNS) metastases and/or leptomeningeal disease requiring immediate treatment with radiation therapy or steroids.
4. Receipt of any cytotoxic chemotherapy within 14 days prior to the first dose of study drugs.
5. QTcF interval >480 msec at Screening (confirmed in triplicate). For patients with ventricular pacemakers, QTcF >500 msec.
6. Known hypersensitivity to carboplatin or other platinum-containing compounds, or mannitol
7. Pregnant or lactating women
8. Prior hematopoietic stem cell or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-05-24 (Actual)

PRIMARY OUTCOMES:
Effect on Overall Survival (OS) | Cohort 1:From date of randomization up to 39 months
  (Cohort 1):To evaluate the effect of trilaciclib on overall survival (OS) compared with placebo in patients receiving first-line gemcitabine and carboplatin.
Effect on Overall Survival (OS) | Cohort 2: From date of randomization up to 28 months
  (Cohort 2): To evaluate the effect of trilaciclib on OS compared with placebo in patients receiving gemcitabine and carboplatin as second-line therapy after treatment with a PD-1/PD-L1 inhibitor in the locally advanced unresectable/metastatic setting

SECONDARY OUTCOMES:
Quality of life/Effects On Chemotherapy-Induced Fatigue | Cycle 1 Day 1 (each cycle is 21 days) up to 14 months
  To assess the effect of trilaciclib on patients' quality of life as measured by time to first confirmed deterioration of fatigue compared with placebo in patients receiving gemcitabine and carboplatin
Myeloprotective Effects | Cycle 1 Day 1 (each cycle is 21 days) up to 14 months
  Occurrence of cytopenias, febrile neutropenia, hospitalization due to chemotherapy-induced myelosuppression, RBC and platelet transfusions, growth factor administration, and dose reductions and delays
Progression Free Survival | From date of randomization up to 14 months)
  To evaluate the effect of trilaciclib on progression-free survival (PFS) compared with placebo in patients receiving gemcitabine and carboplatin.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (71):
- United States (16):
  - Banner M.D. Anderson Cancer Center, Gilbert, Arizona
  - Washington Cancer Institute at MedStar Washington Hospital Center - Oncology Research, Washington D.C., District of Columbia
  - Florida Cancer Specialists - North (SCRI), St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Maryland Oncology Hematology, P.A., Clinton, Maryland
  - Saint Luke's Cancer Specialists, Kansas City, Missouri
  - Comprehensive Cancer Genetics of Nevada, Las Vegas, Nevada
  - Duke Cancer Center, Durham, North Carolina
  - UPC Pinnacle Health Cancer Institute, Pittsburgh, Pennsylvania
  - Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Baptist Cancer Cancer - Oncology, Memphis, Tennessee
  - Tennessee Oncology (SCRI), Nashville, Tennessee
  - Texas Oncology- Austin Central, Austin, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology P.A., Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Peter MacCallum Cancer Centre - Oncology, East Melbourne, Victoria
  - Cabrini Health, Malvern, Victoria
  - Mater Hospital Sydney, North Sydney
- Bulgaria (2):
  - Complex Oncology Center - Burgas, Burgas
  - Medical Ctr Nadezhda Clinical, Sofia
- China (11):
  - Cancer Hospital Chinese Academy of Medical Sciences, Chaoyang, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Yuzhong, Chongqing Municipality
  - Sun Yat-sen University Cancer Center, Yuexiucun, Guangzhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Anhui Provincial Hospital, Harbin, Heilongjiang
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Fudan University Shanghai Cancer Center, Shanghai
- France (6):
  - Centre Jean Bernard, Le Mans, Europe
  - Centre Francois Baclesse, Caen
  - ICM-Val d'Aurelle, Montpellier
  - Centre Hospitalier de Poitiers, Poitiers
  - Pharmacie Essais Cliniques, Toulouse
  - Centre Leon Berard, Villejuif
- Georgia (7):
  - High Technology Hospital MedCenter LTD, Batumi, Adjara
  - Acad.Fridon Todua Medical Center - Research Institute of Clinical Medicine, Tbilisi
  - ARENSIA Exploratory Medicine Harmony Health, Tbilisi
  - LTD Israeli-Georgian Medical Research Clinic Helsicore, Tbilisi
  - LTD Multiprofile Clinic Consilium Medulla, Tbilisi
  - TIM - Tbilisi Institute of Medicine LTD, Tbilisi
  - Institute Of Clinical Oncology LTD, Tbilisi
- IMSP Institutul Oncologic, ARENSIA Exploratory Medicine, Chisinau, Moldova
- Poland (6):
  - Med-Polonia Sp. Z o.o., Poznan, Greater Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Instytut MSF Sp. z. o.o., Lodz
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Oddzial Chorob Rozrostowych, Lodz
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej - Curie - Panstwowy Instytut Badawczy, Warsaw
- Russia (5):
  - Saint-Petersburg State Budgetary Healthcare Institution "City Clinical Oncology Dispensary", Moscow, Balashikha
  - SAHI Republcx Clinical Oncology Dispensary of the Ministry of Healthcare of Tatarstan Republix, Kazan'
  - FSBI Russian Scientific Center of Roentgenoradiology of the MoH of Russia, Moscow
  - State Budgetary Healthcare Institution of Moscow Region "Moscow Reginoal Oncology Dispensary", Moscow
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncological Dispensary", Omsk
- Spain (7):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Puerta de Hierro Majadahonda, Madrid, Majadahonda
  - Hospital Universitario de Badajos, Badajoz
  - Hospital Universitario 12 de Octubre, Barcelona
  - Vall d'Hebrón University Hospital, Barcelona
  - Hospital Clìnic de Barcelona, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
- Ukraine (5):
  - Yuri Prokopovich Spizhenko, Kapitanivka, Kyivska Oblast
  - Komunalne nekomertsiine pidpryiemstvo Sumskoi oblasnoi rady Sumskyi oblasnyi onkolohichnyi dyspanser, Sumy, Sumska Oblast
  - Komunalne nekomertsiine pidpryiemstvo Ternopilskyi oblasnyi klinichnyi onkolohichnyi dyspanser Ternopilskoi oblasnoi rady, Ternopil, Ternopil Oblast
  - Volynskyi oblasnyi medychnyi tsentr onkolohii, Lutsk, Volyn Oblast
  - Komunalne nekomertsiine pidpryiemstvo Miska klinichna likarnia No 4 Dniprovskoi miskoi rady, Dnipro

REFERENCES:
- [Derived] Goel S, Tan AR, Rugo HS, Aftimos P, Andric Z, Beelen A, Zhang J, Yi JS, Malik R, O'Shaughnessy J. Trilaciclib prior to gemcitabine plus carboplatin for metastatic triple-negative breast cancer: phase III PRESERVE 2. Future Oncol. 2022 Oct;18(33):3701-3711. doi: 10.2217/fon-2022-0773. Epub 2022 Sep 22. PMID 36135712